CLINICAL TRIAL: NCT03893097
Title: A Proof-of-concept Trial to Evaluate Artesunate-mefloquine as a Novel Alternative Treatment for Schistosomiasis in African Children
Brief Title: Evaluation of Artesunate-mefloquine as a Novel Alternative Treatment for Schistosomiasis in African Children
Acronym: SchistoSAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Institut de Recherche en Santé, de Surveillance Épidémiologique et de Formation (IRESSEF) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1269/18
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Schistosoma Haematobium; Schistosoma Mansoni
Keywords: Schistosoma; Schistosomiasis; Senegal; Praziquantel; Artesunate; Mefloquine
MeSH Terms: conditions — Schistosomiasis haematobia; Schistosomiasis | interventions — Praziquantel; Artesunate; Mefloquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Praziquantel (Active Comparator): Participants in this arm will receive one dose of PZQ at baseline at 40 mg/kg.
  Interventions: Drug: Praziquantel
- Artesunate-Mefloquine (Experimental): Participants in this arm will receive the Artesunate-Mefloquine (fixed-drug)combination at 4 mg/kg artesunate and 8 mg/kg mefloquine at 3 consecutive days. This will be repeated twice; at week 6 and week 12.
  Interventions: Drug: Artesunate + Mefloquine

INTERVENTIONS:
Drug: Praziquantel — 40 mg/kg at baseline
  Arms: Praziquantel
Drug: Artesunate + Mefloquine — 4mg/kg artesunate and 8 mg/kg mefloquine at baseline (3 consecutive days) and repeated at Week 6 and Week 12
  Arms: Artesunate-Mefloquine

SUMMARY:
The SchistoSAM study is an open label, two-arm, individually-randomized controlled trial with a non-inferiority design, conducted in northern Senegal.

The study aims at determining if the efficacy of one and of repeated courses of artesunate-mefloquine (AM) is respectively similar to or higher than that of a standard praziquantel (PZQ) treatment. Secondly, the study will assess if novel DNA- and antigen-based diagnostics are more accurate than microscopy in assessing antischistosomal treatment response.

DETAILED DESCRIPTION:
The SchistoSAM study is an open label, two-arm, individually-randomized controlled trial with a non-inferiority design, conducted in northern Senegal.

The study aims at determining if the efficacy of one and of repeated courses of artesunate-mefloquine (AM) is respectively similar to or higher than that of a standard praziquantel (PZQ) treatment. Secondly, the study will assess if novel DNA- and antigen-based diagnostics are more accurate than microscopy in assessing antischistosomal treatment response.

For this purpose, 726 school children, aged 6-14 years old and infected with Schistosoma (as demonstrated by presence of eggs in stool and/or urine) will be randomized in one of the following arms:

1. AM, available in fixed dose tablets of 25/50 mg and 100/200 mg will be administered once daily for three days in a dose closest to 4 mg/kg artesunate and 8 mg/kg mefloquine. This treatment course will be repeated 2 times at 6-week intervals.
2. PZQ, available in tablets of 600 mg, will be administered as a single dose of 40 mg/kg.

Trial participants will be regularly followed-up:

1. At each dose administration
2. At day 7 after each dose for follow-up of safety
3. At week 4, 10 and 16 for parasitological assessment and follow-up of safety
4. At week 6 and 12 for clinical assessment before the second and third drug administration (only in the AM arm)
5. At week 24 and 48 for assessment of Schistosoma spp. and malaria infection and associated morbidity (compared to baseline)

ELIGIBILITY:
Inclusion Criteria:

1. Children ≥6 and ≤14 years of age
2. Enrolled in one of the selected primary schools in the region
3. Infected with schistosomiasis (i.e. Schistosoma spp. eggs in urine and/or stool)
4. Informed consent from parents/guardians signed

Exclusion Criteria:

1. History of, or ongoing, epilepsy or psychiatric illness (I.e. recent history of depression, generalized anxiety disorder; history of psychosis, schizophrenia or other major psychiatric disorders) or known hypersensitivity to one of the three study drugs
2. Chronic medication for any reason
3. Any severe underlying illness, including severe malnutrition or severe chronic schistosomiasis, based on clinical judgement
4. Any febrile illness
5. Exposure to PZQ or ACT within the three previous months.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 726 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of a single course of artesunate-mefloquine for the treatment of schistosomiasis, compared to the standard PZQ regimen: Parasitological cure rate | Week 4
  Parasitological cure rate, as assessed by microscopy, after administration of PZQ and after one AM course
Number of safety events of a single course of artesunate-mefloquine for the treatment of schistosomiasis, compared to the standard PZQ regimen | Week 4
  Frequency of drug-related adverse events and serious adverse events
Number of safety events of a single course of artesunate-mefloquine for the treatment of schistosomiasis, compared to the standard PZQ regimen | Week 4
  Pattern of drug-related adverse events and serious adverse events

SECONDARY OUTCOMES:
Evaluate the cumulative efficacy of two additional courses of AM (at 6-week intervals each) for the treatment of schistosomiasis, compared to a single course of AM, and compared to the standard regimen: Cure rate | Week 48
  Cure rate, as assessed by microscopy, after the second and after the third AM administration
Number of safety events of two additional courses of AM (at 6-week intervals each) for the treatment of schistosomiasis, compared to a single course of AM, and compared to the standard regimen. | Week 16
  Frequency of adverse events and serious adverse events up to 4 weeks after the second and third AM administration.
Determine the egg reduction rate obtained after single and repeated courses of AM compared to the standard PZQ regimen. | Week 48
  Egg reduction rate after administration of PZQ and after each AM course
Determine the parasitological efficacy of single and repeated courses of AM by Schistosoma species and by infection intensity. | Week 16
  Cure rate and egg reduction rate by Schistosoma species (S. haematobium and S. mansoni) and by initial Schistosoma infection intensity after PZQ administration and single and repeated courses of AM
Assess the impact of repeated AM courses on schistosomiasis-related morbidity | Week 48
  Prevalence and severity of general and organ-specific schistosomiasis morbidity (as assessed by clinical evaluation, ultrasound, point-of-care morbidity markers and hemoglobin level) compared to baseline and compared to the control arm.
Determine the diagnostic accuracy of novel schistosomiasis antigen- and DNA-based diagnostic assays to monitor antischistosomal treatment response | Week 48
  Diagnostic accuracy of the different conventional and novel diagnostic tests (antigen- and DNA-based) at baseline and at defined time points after treatment compared to conventional stool/urine microscopy, and to composite reference standards (any positive test would be considered as infection).
Determine the effect of repeated AM courses on prevalence of P. falciparum infection as well as on incidence and morbidity of clinical malaria in school-age children with schistosomiasis | Week 48
  * Prevalence of malaria infection, as assessed by molecular testing of dried blood spots.
  * Incidence of clinical malaria, as assessed by the number of incident malaria cases diagnosed through passive case detection during the study period (by standard malaria rapid tests and molecular diagnostics on dried blood spots).
  * Frequency and severity of anemia, as assessed by determination of hemoglobin levels.
Monitor the prevalence of Pf molecular markers associated with mefloquine resistance and the potential emergence of reduced artesunate susceptibility | Week 48
  Prevalence and patterns of mutations in the K13 gene (for artemisinin susceptibility) and increased copy number of the Pfmdr1 gene or other relevant mutations (for mefloquine resistance) observed in the molecular surveys Presence and patterns of mutations observed in incident malaria cases.
Number of safety events of two additional courses of AM (at 6-week intervals each) for the treatment of schistosomiasis, compared to a single course of AM, and compared to the standard regimen. | Week 16
  Pattern of adverse events and serious adverse events up to 4 weeks after the second and third AM administration.

CONTACTS AND LOCATIONS:
Overall Officials: Moustapha Mbow, MD, Principal Investigator — IRESSEF
Locations (1):
- Institut de Recherche en Santé, de Surveillance Épidémiologique et de Formation (IRESSEF), Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from 726 subjects, infected with Schistosomiasis and treated according to protocol in one of two arms. The final dataset will include phenotypic data such as demographics and medical history, results of the different diagnostic tests under investigation, clinical signs and symptoms, echography findings on Schistosomiasis induced morbidity, results of indirect morbidity markers under investigation, presence or absence of Plasmodium falciparum (Pf) and of Pf molecular resistance markers. All the individual participant data and additional supporting information will be deposited, after deidentification, at the IDDO - Schistosomiasis/STHs Data Platform. This is a platform specifically for Schistosomiasis/STHs data and is part of the IDDO project, an international collaboration hosted by the University of Oxford. The repository has data access policies and procedures consistent with ITM data sharing policies.
Supporting Information: Study Protocol, ICF
Time Frame: We anticipate to deposit the individual participant data into the IDDO repository as soon as possible after publication of both findings on treatment efficacy and diagnostic accuracy, but no later than within one year. No end date is established for availability and access to the submitted data.
Access Criteria: For the first five years from submission of the data, decisions regarding data access for third parties will be taken by the authors in collaboration with the ITM Data Access Committee (DAC). After five years, all requests for access to the Data from third parties shall automatically be delegated to DAC of IDDO. The IDDO DAC will provide controlled access to third party researchers whose applications for Data held within the IDDO repository are approved by the DAC in accordance with specific Data Access Guidelines.
  All requests are reviewed for qualifications of the researchers, the design and objectives of the secondary research, analysis plan and publication plan, consistency with ITM data sharing policies, applicable laws and regulations, and required ethics approvals.
URL: http://www.itg.be/E/data-sharing-open-access

REFERENCES:
- [Derived] Bottieau E, Mbow M, Brosius I, Roucher C, Gueye CT, Mbodj OT, Faye BT, De Hondt A, Smekens B, Arango D, Burm C, Tsoumanis A, Paredis L, Van Herrewege Y, Potters I, Richter J, Rosanas-Urgell A, Cisse B, Mboup S, Polman K. Antimalarial artesunate-mefloquine versus praziquantel in African children with schistosomiasis: an open-label, randomized controlled trial. Nat Med. 2024 Jan;30(1):130-137. doi: 10.1038/s41591-023-02719-4. Epub 2024 Jan 4. PMID 38177851
- [Derived] Roucher C, Brosius I, Mbow M, Faye BT, De Hondt A, Smekens B, Arango D, Burm C, Tsoumanis A, Paredis L, van Herrewege Y, Potters I, Cisse B, Mboup S, Polman K, Bottieau E. Evaluation of Artesunate-mefloquine as a Novel Alternative Treatment for Schistosomiasis in African Children (SchistoSAM): protocol of a proof-of-concept, open-label, two-arm, individually-randomised controlled trial. BMJ Open. 2021 Jun 24;11(6):e047147. doi: 10.1136/bmjopen-2020-047147. PMID 34168029